CLINICAL TRIAL: NCT06545383
Title: The Effect of Dynamic Neuromuscular Stabilization Exercises on Balance, Proprioception and Functional Level in Patients With Lower Extremity Lymphedema
Brief Title: The Effect of Dynamic Neuromuscular Stabilization Exercises in Patients With Lower Extremity Lymphedema
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Büşra Çiftçi, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUC-FTR-BC-01
Record Dates: First submitted 2024-07-04; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Lymphedema, Lower Limb
Keywords: Lower Extremity Lymphedema; Exercise
MeSH Terms: conditions — Lymphedema; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Comparing two exercise groups
Who Masked: Participant
Masking Description: the participant will not know which exercise group she/he is in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic Neuromuscular Stabilization Exercises (Experimental): Participants will be taught face-to-face the same home exercise program that was taught to the Exercise Group. In addition, Dynamic Neuromuscular Stabilization (DNS) exercises will be performed. Participants will be informed about DNS exercises and postures. Progress will be made in the exercises step by step. The exercises performed during the positions will be increased by performing 3 sets of 10 repetitions in the first 3 weeks and 3 sets of 15 repetitions in the last 3 weeks.
  Interventions: Other: Dynamic Neuromuscular Stabilization Exercises
- Exercise (Active Comparator): Participants will be taught the home exercise program face to face. Exercises will start with diaphragmatic breathing. Breathing exercises will be done in 2 sets of 10 repetitions. Lower extremity joint range of motion exercises; It will consist of hip flexion in the supine position, hip abduction in the side lying position, hip extension and knee flexion in the prone position, knee extension and ankle dorsi-plantar flexion in the sitting position. Exercises will be increased to 3 sets of 10 repetitions for the first 3 weeks, and 3 sets of 15 repetitions after the 3rd week. After the exercises, they will be asked to walk for 20 minutes at moderate intensity on a flat surface. Additionally, the control group will be asked to walk at moderate intensity.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Dynamic Neuromuscular Stabilization Exercises — Exercises will last 45 minutes and will be 3 days a week for 6 weeks. Additionally DNS exercises will be performed in 40-minute sessions, 2 days a week for 6 weeks.
  Arms: Dynamic Neuromuscular Stabilization Exercises
Other: Exercise — Exercises will last 45 minutes and will be 3 days a week for 6 weeks. Additionally, the control group will be asked to walk at moderate intensity for 40 minutes, 2 days a week, for 6 weeks.
  Arms: Exercise

SUMMARY:
After lower extremity lymphedema, individuals physical activity levels and functionality remain very low. This decrease can cause balance problems over time. Surgical and medical treatments reduce the nerve conduction efficiency of the nervous system and negatively affect proprioception, which is the perception of the joint's position in space during movement. Increasing errors in joint position sense reduce control of movement and restrict active movement, which lead to an assumption that balance could be affected. Joint position sense and balance may be negatively affected, causing injuries, and injuries may cause damage to ligaments and sensory nerve fibers. The main aim of the Dynamic Neuromuscular Stabilization (DNS) approach is to restore physiological movement patterns. By activating the deep stabilizer system with DNS exercises, joint movements could improved, and exercise positions will have positive effects on the quality of sensory perception. In addition, positive effects on balance are expected due to decrease in joint position sense errors. Therefore, the aim of the study is to investigate/understand the effect of DNS exercises on balance, proprioception and functional level in patients with lower extremity lymphedema. This study will provide information for researchers, therapists, and patients by determining the effectiveness of DNS exercises in patients with lower extremity lymphedema.

from Bezmiâlem Vakıf University Faculty of Medicine, Department of Physical Therapy and Rehabilitation, who have been diagnosed with lymphedema due to primary or secondary causes and have progressed to the Complex Decongestive Treatment Phase 2, will constitute the population of the study. The study will be carried out at Istanbul University-Cerrahpaşa Department of Physiotherapy and Rehabilitation.

The study will consist of two groups. Both groups will be included in an exercise program consisting of breathing exercises, active joint range of motion exercises and walking training. Exercises will be given as a home program for 6 weeks, 3 days a week, 45 minutes a day. Additionally, patients in the Control group will be asked to walk for 40 minutes 2 days a week for 6 weeks. In the intervention group, they will additionally be included in a program consisting of individualized DNS exercises for 40 minutes a day, 2 days a week for 6 weeks. All patients will be asked to wear compression garments during exercises.

DETAILED DESCRIPTION:
The study will be carried out with 42 cases referred from Bezmialem Vakif University Faculty of Medicine Hospital Physical Therapy and Rehabilitation Clinic. It will be carried out at Istanbul University-Cerrahpasa Department of Physiotherapy and Rehabilitation. Patients will be randomly divided into Intervention and Control groups. Both groups will be included in an exercise program consisting of breathing exercises that stimulate the lymphatic system in the thoracic region, active joint range of motion exercises and walking training to increase muscle strength and endurance. Exercises will be given as a home program for 6 weeks, 3 days a week, 45 minutes a day. Additionally, patients in the Control Group will be asked to walk for 40 minutes 2 days a week for 6 weeks. In the Intervention Group, they will additionally be included in a program consisting of different postural positions and individualized Dynamic Neuromuscular Stabilization (DNS) exercises added while maintaining the position, 2 days a week, 40 minutes a day for 6 weeks. All patients will be asked to wear compression garments during exercises. Patients' demographic information (age, height, weight, dominant extremity, occupation and education level), duration (years) and stage of lymphedema complaints, and medical history (chemotherapy, radiotherapy and surgical treatment) will be questioned. Participants' lower extremity edema will be evaluated with a tape measure. Their static balance will be evaluated by the one-leg standing test, their dynamic balance by the Y balance test, and their proprioception sense by the joint position sense test. The functional levels of the patients will be evaluated using the 10-meter walk test and the 'Lower Extremity Functional Scale'. Additionally, individuals' fear of falling will be questioned with the 'International Fall Activity Scale'. All evaluations will be made before treatment and after the 6th week of treatment is completed. The sample size was calculated with the G* Power 3.1 power analysis program. Considering the effect size of edema evaluation, which is one of the outcome measurements, as 0.90, the sample size required for a 95% study power was calculated with a 95% confidence interval. It was determined that the number of cases to be included in each group was at least 19. In order to preserve the 95% study power against the possibility of cases falling out of the study, 21 cases will be included by adding a 10% drop margin to each group. Statistical analysis of the data obtained from the study "Statistical Package for Social Sciences" (SPSS) Version 22.0 (SPSS inc., Chicago, USA) statistical program. Whether the data conforms to normal distribution will be determined by the " Shapiro-Wilk Test". According to the analysis results of this test, parametric tests will be applied in the analysis of data that conforms to normal distribution, and non -parametric tests will be applied in the analysis of data that does not comply with normal distribution. In the statistical analysis of the study, the variables evaluated will be defined with mean (Mean), standard deviation (SD) and percentage (%) values. For quantitative/numerical data comparing the demographic and clinical characteristics of the groups that make up the study, Independent Samples T-test and Chi-square test will be used for qualitative/non-numerical data. Results will be considered significant at the 95% confidence interval and significance level of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Being diagnosed with lymphedema due to primary or secondary causes in the lower extremity
* Having progressed to Complex Decongestive Treatment Phase 2
* Volunteering to participate in research

Exclusion Criteria:

* No mental or cognitive problems
* Not receiving any other concurrent conservative or surgical treatment during the study.
* Presence of metastatic cancer
* Having a neurological disorder that may affect balance or an orthopedic disorder that may prevent walking
* Presence of active infection in the affected limb
* Uncontrolled hypertension, presence of serious cardiovascular system disease
* There is a risk of deep vein thrombosis
* Presence of open skin wound
* Having a history of falling in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Static Balance on the One-Leg Stance Test | Six week
  With this test, static balance is evaluated. It correlates well with other balance tests. It is time efficient and does not require the use of special equipment. The test is performed without shoes on a smooth and hard surface. It is measured how long the individual can stand on one leg without assistance, with the arms close to the body. The time is recorded with chronometer. The duration starts when the patient lifts his foot off the ground and ends when his foot touches the ground. The test ends when the foot is moved or the time reaches a maximum of 60 seconds. The average of 3 repetitions is taken. The time is recorded in seconds. Standing on one leg for longer periods of time indicates better balance. The test will be applied with eyes open and closed.
Change from Baseline in Dynamic Balance on the Y Balance Test | Six week
  The Y balance test evaluates the dynamic balance of the lower extremity. Three lines in the shape of a "Y" are drawn in the test area, with a 135-degree angle between the back strips and the front strip and a 45-degree angle between the back strips. The patient is asked to place his foot on the side to be tested at the intersection of the lines. The patient gently touches the anterior, posteriolateral, posteromedial directions with the other foot and brings it back to the fixed leg. During this time, care is taken not to lift the heel of the other foot. If the balance is disrupted, the test is canceled and repeated. The point where the foot touches is marked and the distance to the intersection point is recorded in centimeters. The test is repeated 3 times and the average is recorded.

SECONDARY OUTCOMES:
Change from Baseline in Proprioception on the Joint Position Sense Test | Six week
  Digital inclinometer; It is a device that is simple to use, affordable, portable, and makes quick measurements compared to expensive and complex equipment. Joint position sense is evaluated by the patient actively moving the extremity to the specified angle. The digital inclinometer is fixed on the limb using a strap. The patients' full range of motion in the joint to be evaluated is measured and 50% of these angles are selected as the target position. The therapist brings the person to the target position and asks him to stop there for 5 seconds and focus on the point he is in, then return to the starting position. This movement is repeated 3 times for the patient to learn the position. During the test, the participants' eyes are covered with an eye patch. Testing is performed when participants actively reposition the joint to the target position. When the participant feels that he/she has reached the target position, he/she stops and the test ends in the position where he/she stands
Change from Baseline in Functional Level on the 10 Meters Walking Test | Six week
  The starting and finishing lines are determined in the 10 meter long test area. The time started when the participant walking at his own pace is at the starting line and ends at the finish line. The average value of three measurements is recorded in meters per second (m/s).
Change from Baseline in Functional Level on the Lower Extremity Functional Scale | Six week
  The Lower Extremity Functional scale, which evaluates the functional level of individuals, consists of 20 questions. The Turkish validity and reliability of the scale was determined by Citaker et al. Answers to the questions; 0: Extreme difficulty or inability to perform the activity, 1: A great deal of difficulty, 2: Moderate difficulty, 3: Some difficulty, 4: No difficulty at all. An increase in the score indicates a better functional level.
Change from Baseline in Edema on the Environmental Measurement Methods | Six week
  Edema is evaluated based on certain reference points. Although it varies among clinicians, it is easy to use and common in the clinic. It is recommended that measurements be made by the same therapist. In a long sitting position, when the ankle is neutral, measurements are made with a tape measure at 5 centimeter intervals, using the malleolus as a reference. The volume is determined using the truncated cone formula with the obtained values. Frustum formula; V= [h x (R1²+R1.R2+R2²)] / (12 x π), Total Leg Volume=V1+V2+V3…+Vn (V: Volume of each conical segment, h: Range used in environmental measurement, R1: Base circumferential measurement of tapered segment, R2: Upper circumferential measurement of tapered segment, n: Number of conical segments).
Change from Baseline in Fear of Falling on the Falls Efficacy Scale International (FES-I) | 6 week
  The Falls Efficacy Scale International assesses anxiety about the possibility of falling through activities. The Turkish validity and reliability study of the scale was conducted by Ulus et al. It was conducted by in 2012. The scale consists of 16 questions and is answered as 'I never worry (1 point)', 'I worry a little (2 points)', 'I worry quite a bit (3 points)' and 'I worry a lot (4 points)'. The total score is recorded, an increase in the score indicates an increase in the fear of falling.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Çiftçi, BSc, Principal Investigator — Istanbul University - Cerrahpasa; Rüstem Mustafaoğlu, Assoc Prof D, Principal Investigator — Istanbul University - Cerrahpasa; Teoman Aydın, Prof Dr, Principal Investigator — Bezmialem Vakif University
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University-Cerrahpasa, Istanbul, Büyükçekmece
  - Bezmialem Vakif University, Istanbul, Fatih

IPD SHARING:
Plan to Share IPD: No